CLINICAL TRIAL: NCT01313598
Title: An Open-label, Dose Escalating Phase Ib Study for the Assessment of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Intravenous Doses of GLPG0187 in Subjects With Solid Tumors
Brief Title: GLPG0187: Safety, Tolerability and Pharmacokinetics in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLPG0187-CL-102; 2010-021164-15 (EudraCT Number)
Record Dates: First submitted 2011-02-28; First posted 2011-03-14 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Solid Tumors
Keywords: Patients with solid tumors; Treatment-refractory
MeSH Terms: interventions — GLPG0187

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GLPG0187 (Experimental): GLPG0187 for infusion
  Interventions: Drug: GLPG0187

INTERVENTIONS:
Drug: GLPG0187 — continuous IV infusion

SUMMARY:
The purpose of the study is to determine the safety and tolerability of GLPG0187 administered through continuous intravenous infusion and to explore its preliminary clinical efficacy in patients with solid tumors.

DETAILED DESCRIPTION:
Patients with pathologically confirmed diagnosis of advanced, recurrent, or metastatic cancer and who are refractory to standard therapy or for whom no standard therapy exists will first receive a one-hour infusion of a defined dose of GLPG0187. If well tolerated, one week later a three-week continuous infusion is started. If according to the investigator a subject has a clinical benefit from treatment with GLPG0187, the treatment cycle may be repeated until disease progression, Dose Limiting Toxicity (DLT), or the patient chooses to stop or cannot/will not comply with study procedures.

Throughout treatment, safety and tolerability will be monitored. Within one patient, a fixed dose (infusion rate) will be used. If at a given dose-level sufficient patients have been treated without reaching DLT, the dose for the next group of patients will be increased. This can be repeated until DLT is established, or the scheduled maximum dosage is reached.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of advanced, recurrent, or metastatic cancer who are refractory to standard therapy or for whom no standard therapy exist.
* Age of 18 years or older.
* Measurable (according to RECIST 1.1) and evaluable disease as determined by the Investigator.
* ECOG Performance Status ≤ 2.
* Estimated life expectancy of at least 12 weeks.
* Toxicities incurred as a result of previous anticancer therapy (radiation therapy, chemotherapy, or surgery) must be resolved to ≤ Grade 2.
* Written informed consent according to local guidelines.

Exclusion Criteria:

* Prior Treatment:

  * Less than 4 weeks since the last treatment with other cancer therapies, (i.e. endocrine therapy, immunotherapy, chemotherapy, etc.), and < 6 weeks for nitrosoureas and Mitomycin C.
  * Prior therapy with integrin receptor antagonists
* Current Treatment:

  * Chronic daily treatment with corticosteroids (dose of 10 mg/day or more methylprednisolone or equivalent), with the exception of inhaled steroids.
  * Current or recent (within 30 days of first study treatment) treatment with another investigational drug or participation in another investigational study.
* Hematology, coagulation and biochemistry:

  * Inadequate bone marrow function: Absolute Neutrophil Count (ANC): < 1.5 x 10E9/L, or platelet count <100 x 10E9/L or hemoglobin < 6 mmol/L.
  * Inadequate liver function, defined as:

    * Serum (total) bilirubin > 2 x the Upper Limit of Normal (ULN) for the institution;
    * Aspartate Amino Transferase (ASAT) or Alanine Amino Transferase (ALAT) > 2.5 x ULN (> 5 x ULN in subjects with liver metastases);
    * Alkaline phosphatase levels > 2.5 x ULN (> 5 x ULN in subjects with liver metastases, or > 10 x ULN in subjects with bone metastases).
  * Inadequate renal function, defined as:

    * Serum creatinine > 1.5 x ULN
    * Urine dipstick for proteinuria > 2+.
* Other:

  * Clinically symptomatic or progressive brain metastases
  * Clinical Leptomeningeal metastases
  * Pregnancy or lactation. Serum pregnancy test to be assessed within 7 days prior to study treatment start, or within 14 days with a confirmatory urine pregnancy test within 7 days prior to study treatment start.
  * For women of childbearing potential (defined as <2 years after last menstruation and not surgically sterile): absence of effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal gel).
  * Major surgical procedure (including open biopsy, excluding central line IV and portacath) within 28 days prior to the first study treatment, or anticipation of the need for major surgery during the course of the study treatment.
  * Congestive heart failure NYHA Class III and IV. Cardiac arrhythmias (except for atrioventricular block type I, Mobitz type, and II, Wenckebach type) signs and symptoms of relevant cardiovascular disease.
  * Known hypersensitivity to any of the study drugs or excipients.
  * Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, physical examination or laboratory findings) that may interfere with the planned treatment, affect subject compliance or place the subject at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Four weeks + three-week cycles
  Patients will be monitored for cardiovascular safety (ECG) and adverse events, and blood- and urine-samples taken before and at fixed timepoints after a one-hour infusion of GLPG0187; if patients tolerate the treatment well, procedures will be repeated before and at fixed timepoints after the start of a three-week continuous infusion patients. Through monitoring and analysis of the blood- and urine-samples, it will be established whether the study medication would have any negative effects on the patient's general condition. Results will indicate whether DLT has occurred.

SECONDARY OUTCOMES:
Pharmacokinetics of GLPG0187 after intravenous infusion. | Up to four weeks.
  Blood samples will be taken at regular timepoints before and on fixed timepoints after start of the one-hour infusion, as well as before and on fixed timepoints during the (first) three-week infusion, to establish the concentration of the study medication in the blood.
Pharmacodynamics of GLPG0187 | Up to four weeks
  Blood samples will be taken at regular timepoints before and on fixed timepoints after start of the one-hour infusion, as well as before and on fixed timepoints during the (first) three-week infusion, to measure the levels of CTx (collagen telopeptide, a bone resorption biomarker).
Preliminary efficacy of GLPG0187 in terms of clinical activity. | Four weeks + three-week cycles
  evaluation of antitumor effects according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Giocondo Lorenzon, MSc, Study Director — Galapagos SASU
Locations (2):
- Netherlands (2):
  - Nationaal Kanker Instituut (NKI), Amsterdam
  - Universitair Medisch Centrum, Utrecht